CLINICAL TRIAL: NCT06476795
Title: The Influence of Chardonnay Marc Intake on Gut and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2034985
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Adiposity; Cardiometabolic Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: We will use a two-arm escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chardonnay Marc Intake Level 1 (Experimental): Daily intake of Chardonnay marc at 1.5 g
  Interventions: Other: Chardonnay Marc
- Chardonnay Marc Intake Level 2 (Experimental): Daily intake of Chardonnay marc at 4.5 g
  Interventions: Other: Chardonnay Marc

INTERVENTIONS:
Other: Chardonnay Marc — Food product made from Chardonnay wine grapes

SUMMARY:
Recently a dietary recommendation of 400 - 600 mg/ day has been proposed for the reduced risk of developing cardiovascular disease. Dietary flavanols can be obtained from the intake of foods such as tea, cocoa, wine, berries and apples. Incorporating Chardonnay Marc (the skins and seeds of Chardonnay grapes) into the diet can be an additional source of dietary flavanols. Like other flavanol-rich foods, Chardonnay Marc provides fiber and polysaccharides that may benefit gut health. This study seeks pilot data on the impact of the daily incorporation of Chardonnay Marc powder into the diet on markers of gut and cardiometabolic health.

DETAILED DESCRIPTION:
The overall study objective is to obtain data on the impact of the dietary incorporation of Chardonnay marc on measures of gut and cardiometabolic health. Towards this goal, an escalation design will be employed to examine the effects of 6 - 12 weeks of daily Chardonnay marc intake on markers of gut permeability, inflammation and cardiometabolic health in obese individuals. Study procedures will be performed during 3 study visits conducted at baseline, and after 6 and 12 weeks of Chardonnay Marc intake. For each study visit, 50 ml of blood (~3.5 tbsp) will be collected. For the first six weeks of the study, the participants will be asked to incorporate 1.5 g of Chardonnay Marc into their diet between the hours of 11 am and 4 pm every day. This level of intake will be increased to 4.5 g of Chardonnay marc everyday from weeks 6-12. Therefore, all individuals will consume Chardonnay marc for at least 12 weeks. The participants will be instructed to not cook or add the Chardonnay Marc to hot foods, however, they will be allowed to add the Marc to tepid or warm foods and beverages. They will also be asked to log their intake and how they incorporated the Marc into their diet via a log.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female, with a cessation of menses for at least 2 years
* 45-70 years of age
* BMI 25- 49.9 kg/m2
* Fasting triglycerides > 120 mg/dL
* Subject is willing and able to comply with the study protocols and procedures.

Exclusion Criteria:

* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Prescription medications and supplements, except for a 6 month stable dose of thyroid medications
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Fruit consumption ≥ 3 cups/day
* Vegetable consumption ≥ 4 cups/day
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke, diabetes
* Peripheral artery disease Raynaud's syndrome or disease
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Self-reported cancer within past 5 years
* Self-reported gastrointestinal disorders, apart from appendix removal
* Unwillingness to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements six weeks prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* All forms of smoking (e.g. vaping, cigarette, cannabis)
* Current enrollee in a clinical research study.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Microvascular function | 12 weeks
  Microvascular function measured by peripheral arterial tonometry

SECONDARY OUTCOMES:
Plasma Cholesterol | 12 weeks
  Circulating levels of plasma lipids
Cytokines | 12 weeks
  Pro-inflammatory Th17 cytokines
short chain fatty acids | 12 weeks
  Plasma and fecal levels of short chain fatty acids
plasma bile acids | 12 weeks
  Circulating levels of primary and secondary bile acids
blood glucose | 12 weeks
  fasting levels of blood glucose
Gene expression | 12 weeks
  gene expression from whole blood
insulin | 12 weeks
  plasma insulin levels after an overnight fast
zonulin | 12 weeks
  serum and fecal zonulin as a measure of gut permeability
lipopolysaccharide binding protein | 12 weeks
  serum measure of gut permeability
Metabolomics | 12 weeks
  plasma levels of untargeted metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No